CLINICAL TRIAL: NCT02537678
Title: Stepped Care for Children After Trauma: Optimizing Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH107522-01 (NIH)
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2019-04

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Care TF-CBT (Experimental): Stepped Care TF-CBT consist of two steps. Step One is a parent-led therapist-assisted treatment and Step Two is standard TF-CBT.
  Interventions: Behavioral: Stepped Care TF-CBT
- Standard TF-CBT (Active Comparator): Standard TF-CBT consist of therapist-directly weekly in-office therapy based on the trauma-focused components of TF-CBT.
  Interventions: Behavioral: Standard TF-CBT

INTERVENTIONS:
Behavioral: Stepped Care TF-CBT — Stepped Care TF-CBT: Patients will receive Step One: 3 (1 hr.) in-office therapist-led sessions over 6 weeks, the parent-child workbook (Stepping Together),60, 61 scheduled weekly phone meetings (15 minutes), and information from the Stepping Together website and the National Center for Childhood Traumatic Stress website (via web or paper for those without access). Children who do not meet responder status will receive Step Two: 9 (1.5 hr.) in-office therapist-directed sessions of TF-CBT over 6 to 8 weeks
  Arms: Stepped Care TF-CBT
Behavioral: Standard TF-CBT — Standard TF-CBT: Patients will receive 12 (1.5 hr.) standard weekly in-office therapist-directed sessions (2 additional weeks allow for scheduling difficulty). TF-CBT includes child, parent and conjoint parent-child sessions addressing the 10 core trauma treatment components of TF-CBT (e.g., parenting skills, affect modulation, cognitive coping, trauma narrative, etc.).
  Arms: Standard TF-CBT

SUMMARY:
Children who are exposed to traumatic events are at risk for developing PTSD and other mental health problems. Although effective treatments for childhood PTSD exist, service delivery approaches that are more accessible, efficient, and cost-effective are needed to improve access to evidence-based treatment. The proposed study furthers our pilot work and evaluates an innovative Stepped Care Trauma-Focused Cognitive Behavioral Therapy designed to optimize treatment in community settings and improve the value and efficiency of trauma-focused treatment for children compared to existing approaches, thereby reducing childhood PTSD and related societal impacts and costs.

DETAILED DESCRIPTION:
Approximately 68-80% of youth will experience at least one potentially traumatic event during their childhood with about one third experiencing more than one traumatic event. Exposure to traumatic events markedly elevates the risk of developing posttraumatic stress disorder (PTSD) and associated impairment. Despite advances in effective trauma-focused treatments for children, the lack of efficient, accessible, personalized, and cost-effective trauma treatment for children is a major public health concern. Thus, there is a critical need for interventions to improve efficiency, access, and cost-effectiveness and to offer tailored approaches that meet the unique needs of the child. The present study builds on the investigators NIH-funded pilot work (1R34MH092373-01A1) that developed an innovative Stepped Care Trauma-Focused Cognitive Behavioral Therapy (SC-TF-CBT). The purpose of the proposed study is to examine how to optimize the efficiency (e.g., via matching children to appropriate treatment dosage at baseline, utilizing second-stage tailoring variables, and identifying mechanisms of change) and cost-effectiveness of Stepped Care TF-CBT. The long-term goal is to develop an effective, efficient, accessible, and cost-effective adaptive Stepped Care TF-CBT intervention that can be available to more trauma-exposed children, and to advance knowledge about service delivery approaches that may be applicable to providing treatment for other childhood mental health disorders. The goal of the study is consistent with the strategic objective to "Develop New and Better Interventions that Incorporate the Diverse Needs and Circumstances of People with Mental Illness," and the research priorities that call for trials that foster prescriptive, personalized mental health care, incorporate tailoring variables to match patient interventions, improve access to services, decrease costs of services, and incorporate measures of putative mechanisms of action in trials in "real world" settings. In a randomized clinical trial with 216 children ages 4 to 12 years at community-based agencies, the following aims are proposed:

Aim 1: To examine Stepped Care TF-CBT (e.g., starting with Step One parent-led, therapist-assisted treatment and then either maintenance or Step Two TF-CBT) relative to standard TF-CBT (e.g., therapist-led treatment);

Aim 2: To examine tailoring variables that could be used to individualize (i.e., tailor) the decision of which children should be assigned at baseline to Stepped Care TF-CBT versus standard TF-CBT;

Aim 3: To examine if changes in the potential mechanisms of change variables (e.g., fear arousal, maladaptive cognitions, negative expectancy, and fear toleration) mediate treatment on child PTSD symptoms (PTSS) and impairment;

Aim 4: To examine the economic cost of delivering Stepped Care TF-CBT versus standard TF-CBT. Children with PTSD are at considerable risk for numerous biopsychosocial problems. Without accessible, effective treatment, these problems tend to persist into adulthood. This study will yield clinically important data which will improve the value and efficiency of treatment of children with PTSD, thereby reducing childhood PTSD and related societal impacts and costs.

ELIGIBILITY:
Parent/Guardian-child dyads enrolled.

Inclusion Criteria:

1. Child experienced at least one traumatic event after the age of 36 months
2. Child age 4-6 must meet at least four PTSD symptoms and children age 7 to 12 must meet at least five PTSD symptoms with at least one symptom in re-experiencing or one symptom in avoidance
3. At enrollment, the child must be between 4-12 years of age
4. The parent/guardian must be willing and able to participate in the treatment and complete informed consent

Exclusion Criteria:

1. Psychosis, mental retardation, autism spectrum disorder in the child or any condition that would limit the caregiver's ability to understand CBT and the child's ability to follow instructions
2. Parent has had substance use disorder (SUD) within the past 3 months.
3. Child or parent is suicidal
4. Child or parent is not fluent in English
5. Child is currently taking psychotropic medication and is not on a stable medication regimen for at least 4 weeks prior to admission to the study. For stimulants or benzodiazepines, the medication regimen must be stable for 2 weeks. If appropriate, a delayed entry will be allowed so that once a child is on a stable dosage the child may be enrolled in the study.
6. Child is receiving trauma-focused psychotherapy during study treatment.
7. Parent/caregiver who would be treatment participant was the perpetrator, or the child was perpetrated by a person who still lives in the home
8. Child is having unsupervised face-to-face contact with the identified perpetrator
9. Siblings

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison A Salloum, PhD, Principal Investigator — University of South Florida
Locations (6):
- United States (6):
  - Children's Home Society, Jacksonville, Florida
  - Directions for Living, Largo, Florida
  - Pasco Kids First, New Port Richey, Florida
  - USF St. Petersburg Family Study Center, St. Petersburg, Florida
  - Suncoast Center, Inc, St. Petersburg, Florida
  - Crisis Center of Tampa Bay, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
The data dictionaries for the descriptive and analyzed data were uploaded for the National Institute of Mental Health (NIMH) Data Archive (Salloum C2318).

REFERENCES:
- [Background] Salloum A, Scheeringa MS, Cohen JA, Storch EA. Development of Stepped Care Trauma-Focused Cognitive-Behavioral Therapy for Young Children. Cogn Behav Pract. 2014 Feb 1;21(1):97-108. doi: 10.1016/j.cbpra.2013.07.004. PMID 25411544
- [Background] Salloum A, Scheeringa MS, Cohen JA, Storch EA. Responder Status Criterion for Stepped Care Trauma-Focused Cognitive Behavioral Therapy for Young Children. Child Youth Care Forum. 2015 Feb;44(1):59-78. doi: 10.1007/s10566-014-9270-1. PMID 25663796
- [Result] Salloum A, Robst J, Scheeringa MS, Cohen JA, Wang W, Murphy TK, Tolin DF, Storch EA. Step one within stepped care trauma-focused cognitive behavioral therapy for young children: a pilot study. Child Psychiatry Hum Dev. 2014 Feb;45(1):65-77. doi: 10.1007/s10578-013-0378-6. PMID 23584728
- [Result] Salloum A, Lu Y, Chen H, Quast T, Cohen JA, Scheeringa MS, Salomon K, Storch EA. Stepped Care Versus Standard Care for Children After Trauma: A Randomized Non-Inferiority Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2022 Aug;61(8):1010-1022.e4. doi: 10.1016/j.jaac.2021.12.013. Epub 2022 Jan 12. PMID 35032578
- [Derived] Salloum A, Boedeker P, Morris C, Storch EA. Suicidal Ideation, Clinical Worsening and Outcomes among Child Participants in Trauma-Focused Treatment. Res Child Adolesc Psychopathol. 2025 May;53(5):687-700. doi: 10.1007/s10802-024-01242-5. Epub 2024 Sep 26. PMID 39325087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from six community clinics between October 2015 and April 2019 from five community behavioral health nonprofit organizations and one university community-based clinic. The first participant was enrolled 10/6/2015 and the last participant was enrolled 4/19/2019.
Pre-assignment Details: Parent/guardian-child dyads participated. 212 dyads enrolled. 183 dyads met inclusion and were randomized to treatment. Exclusion before assignment included: Less than 5 trauma symptoms, perpetrator in home, not wanting to participate, no trauma after age 3, cognitive impairment, did not attended assessment, substance abuse within past 3 months, unsupervised visits with perpetrator, medication not stable, no traumatic symptoms, parent suicidal, autism spectrum, parent unable/unwilling.
Groups:
- Stepped Care TF-CBT: Participants (parent-child dyads) received Step One which is a parent-led therapist assisted treatment: 3 therapist-led sessions along with 11 parent-child meetings using a parent-child workbook. Children who do not meet responder status will receive Step Two: 9 therapist-directed sessions of TF-CBT. Two as needed sessions could be provided
- Standard TF-CBT: Participants (parent-child dyads) received therapist led trauma-focused cognitive behavioral therapy (TF-CBT). Two as needed sessions could be provided.
Period: Baseline to Post-treatment
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Started | 91 (91 parents/guardians and 91 children started.) | 92 (92 parents/guardians and 92 children started.)
Completed Post-treatment | 61 (61 parents/guardians and 61 children completed post-treatment.) | 71 (71 parents/guardians and 71 children completed post-treatment.)
Completed | 61 (61 parent/guardian-child dyads completed.) | 71 (71 parent/guardian-child dyads completed.)
Not Completed | 30 | 21
Not completed — Parent/Guardian- child dyads: Never started | 4 | 3
Not completed — Parent/Guardian-child dyads: Withdrew | 4 | 4
Not completed — Parent/Guardian-child dyads: Unknown | 6 | 5
Not completed — Parent/Guardian-child: Dislike therapy | 2 | 3
Not completed — Parent/Guardian barriers: work, moved, homeless, illness, transportation, perpetrator in home | 14 | 6
Period: Post-treatment to 6 Month Assessment
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Started | 61 (61 parents/guardians and 61 children started.) | 71 (71 parents/guardians and 71 children started.)
Completed | 53 (53 parents/guardians and 53 children completed.) | 64 (64 parents/guardians and 64 children completed.)
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 8 | 7
Period: 6 Month to 12 Month Assessment
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Started | 53 (53 parent/guardians and 53 children started.) | 64 (64 parent/guardians and 64 children started.)
Completed | 53 (53 parent/guardians and 53 children completed.) | 63 (63 parent/guardians and 63 children completed.)
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants represent the parent/guardian-child dyads in each arm. There were a total of 91 children and 91 parent/gaurdians analyzed in Stepped Care Trauma-Focused-CBT (TF-CBT). There were a total of 92 children and 92 parent/garudians analyzed in Standard Care Trauma-Focused-CBT (TF-CBT). Thus, the total analyzed was 366.
Groups:
- Stepped Care Trauma Focused-CBT (TF-CBT): Stepped Care TF-CBT consist of two steps. Step One is a parent-led therapist-assisted treatment and Step Two is standard TF-CBT.
  Parent/Guardian-child dyads participated.
  Stepped Care TF-CBT: Stepped Care TF-CBT: Patients will receive Step One: 3 (1 hr.) in-office therapist-led sessions over 6 weeks, the parent-child workbook (Stepping Together), scheduled weekly phone meetings (15 minutes), and information from the Stepping Together website and the National Center for Childhood Traumatic Stress website (via web or paper for those without access). Children who do not meet responder status will receive Step Two: 9 (1.5 hr.) in-office therapist-directed sessions of TF-CBT over 6 to 8 weeks
- Standard Trauma Focused-CBT (TF-CBT): Standard TF-CBT consist of therapist-directly weekly in-office therapy based on the trauma-focused components of TF-CBT.
  Parent/Guardian-child dyads participated.
  Standard TF-CBT: Standard TF-CBT: Patients will receive 12 (1.5 hr.) standard weekly in-office therapist-directed sessions (2 additional weeks allow for scheduling difficulty). TF-CBT includes child, parent and conjoint parent-child sessions addressing the 10 core trauma treatment components of TF-CBT (e.g., parenting skills, affect modulation, cognitive coping, trauma narrative, etc.).
- Total: Total of all reporting groups
Arm/Group | Stepped Care Trauma Focused-CBT (TF-CBT) | Standard Trauma Focused-CBT (TF-CBT) | Total
Number analyzed (Participants) | 91 | 92 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] — Child's age: The evaluator conducting the assessment asked the parent/guardian for the child's age in years and asked for the child's date of birth.
  years | 8.32 (2.39) | 7.46 (2.45) | 7.89 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Child's sex: The evaluator conducting the assessment asked the parent/guardian if their child was male or female.
  Participants
    Female | 48 | 53 | 101
    Male | 43 | 39 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Child's ethnicity: The evaluator conducting the assessment asked the parent/guardian if they considered their child to be Hispanic or Latino or not Hispanic or Latino.
  Participants
    Hispanic or Latino | 26 | 23 | 49
    Not Hispanic or Latino | 65 | 69 | 134
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Child's race: The evaluator conducting the assessment asked the parent/guardian for child's race using the following categories: American Indian or Alaskan Native; Asian; Black or African American; Native Hawaiian or other Pacific Islander; White or more than one race.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 30 | 27 | 57
    White | 46 | 48 | 94
    More than one race | 15 | 16 | 31
    Unknown or Not Reported | 0 | 0 | 0
Parent/Guardian Relationship to the child [Count of Participants; unit: Participants] — Parent/Guardian relationship: The evaluator conducting the assessment asked the parent/guardian for their relationship to the child such as mother, father, grandmother, grandfather or other. The researchers then categorized the reported relationships into 'parent' or 'relative'.
  Participants
    Parent | 80 | 88 | 168
    Relative | 11 | 4 | 15
Parent /Guardian ethnicity [Count of Participants; unit: Participants] — Parent/Guardian ethnicity: The evaluator conducting the assessment asked the parent/guardian if they are Hispanic or Latino or not Hispanic or Latino
  Participants
    Hispanic or Latino | 28 | 14 | 42
    Not Hispanic of Latino | 63 | 78 | 141
Parent/Guardian race [Count of Participants; unit: Participants] — Parent/Guardian race: The evaluator conducting the assessment asked the parent/guardian for their race by reading out the following categories: American Indian or Alaskan Native; Asian; Black or African American; Native Hawaiian or other Pacific Islander; White.
  Participants
    White | 54 | 59 | 113
    Black or African American | 36 | 30 | 66
    American Indian/Alaskan Native | 1 | 1 | 2
    Unknown | 0 | 2 | 2
Household income [Count of Participants; unit: Participants] — Parent/Guardian: The evaluator conducting the assessment asked the parent/guardian for their yearly income giving ranges of 0 to 9,999, 10,000 to 24,999, 25,000 to 34,999, 35,000 to 49,999 or 50,000 and above.
  Participants
    $0 -9,999 | 15 | 17 | 32
    $10,000-24,999 | 13 | 22 | 35
    $25,000-34,999 | 13 | 12 | 25
    $35,000-49,999 | 21 | 16 | 37
    $50,000+ | 29 | 25 | 54
Education levels [Count of Participants; unit: Participants] — Parent/Guardian education: The evaluator conducting the assessment asked the parent/guardian for their highest level of schooling. The researchers then matched the ranges to estimate education categories. The categories were: 9 to 11 years indicated no high school diploma, 12 years indicated high school graduate, 13 to 15 years indicated some college, and 16 or more years indicated college graduate and above.
  Participants
    No high school diploma (9-11yrs) | 7 | 7 | 14
    High school graduate (12 years) | 20 | 16 | 36
    Some college (13-15 years) | 41 | 44 | 85
    College graduate and above (16+ years) | 23 | 25 | 48
Parent/Guardian employed [Count of Participants; unit: Participants] — Parent/Guardian employment status: The evaluator conducting the assessment asked the parent/guardian if they were currently employed with the response option of yes or no.
  Participants
    Employed | 63 | 59 | 122
    Not employed | 28 | 33 | 61
Parent/Guardian with posttraumatic stress disorder [Count of Participants; unit: Participants] — Parent/Guardian: The Structured Clinical Interview for Diagnostic and Statistical Manual-5 research version (First et al., 2015) PTSD module was administered by the evaluator conducting the assessment with the parent/guardian to assess for posttraumatic stress disorder.
  Participants
    Parent/guardian met criteria for PTSD | 45 | 27 | 72
    Parent/guardian did not meet criteria for PTSD | 46 | 65 | 111
Parent/Guardian age [Mean (Standard Deviation); unit: years] — Parent/Guardian age: The evaluator conducting the assessment asked the parent/guardian for their date of birth. The evaluator then used a statistical program to calculate the parent/guardians age by using the date of the assessment and their date of birth.
  years | 38.23 (10.11) | 36.52 (9.97) | 37.37 (10.05)
Parent/Guardian relationship status [Count of Participants; unit: Participants] — Parent/Guardian relationship status: The evaluator conducting the assessment asked the parent/guardian if their current relationship status was single, married, divorced, separated, widowed or other.
  Participants
    Single | 34 | 29 | 63
    Married | 25 | 26 | 51
    Divorced | 12 | 14 | 26
    Separated | 12 | 13 | 25
    Widowed | 3 | 4 | 7
    Other | 5 | 6 | 11
Trauma Symptom Checklist for Young Children Posttraumatic Stress Symptoms [Mean (Standard Deviation); unit: units on a scale] — Child posttraumatic stress: The Trauma Symptom Checklist for Young Children (TSCYC; Briere, 2005) is a caregiver report measure of trauma symptom severity in children ages 3-12 years that includes a 27-item posttraumatic stress symptom total subscale (TSCYC-PTS). The parent/guardian completed this measure using an online program. The range of the TSCYC-PTS is 27 to 108 with higher scores indicating more severe posttraumatic stress symptoms.The change in the TSCYC-PTS will be used to measure change in child's posttraumatic stress symptoms.
  units on a scale | 50.53 (12.15) | 51.34 (13.50) | 50.93 (12.81)
Child Sheehan Disability Scale Parent Version [Mean (Standard Deviation); unit: units on a scale] — Child impairment: The Child Sheehan Disability Scale (Sheehan , 2008) is an adapted caregiver version (Whiteside, 2009) with 5-items to measure childhood impairment. The change in impairment scale will be used to measure change in impairment. Scores range from 0 to 50 with higher scores indicating greater impairment.
  units on a scale | 20.99 (10.80) | 21.29 (12.86) | 21.14 (11.85)

OUTCOME MEASURES:

1. Primary Outcome: Trauma Symptom Checklist for Young Children Posttraumatic Stress Symptoms
Description: Trauma Symptom Children for Young Children Posttraumatic Stress total score will measure changes in child posttraumatic stress symptoms for children ages 4-12. Score ranges from 27 to 108 with higher scores indicating greater posttraumatic stress symptoms.
Time Frame: Post treatment
Population: Intent to treat population (ITT; all participants assigned to stepped care TF-CBT and standard TF-CBT). Multiple imputation was applied for ITT analysis, with ten imputations generated at item level and individual level.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stepped Care TF-CBT: Participants received Step One which is a parent-led therapist assisted treatment: 3 therapist-led sessions along with 11 parent-child meetings using a parent-child workbook. Children who do not meet responder status will receive Step Two: 9 therapist-directed sessions of TF-CBT. Two as needed sessions could be provided
- Standard TF-CBT: Participants received therapist led trauma-focused cognitive behavioral therapy (TF-CBT). Two as needed sessions could be provided.
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 36.00 (10.52) | 35.57 (9.17)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Based on the actual randomization of 183 participants (SC-TF-CBT=91; standard TF-CBT=92), we had more than 80% power to show that SC-TF-CBT is at least as effective as standard TF-CBT with alpha of .05 and a non-inferior margin of 0.41 SD units; Test type: Non-Inferiority — We planned 0.41 standard deviation (SD) as the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied at post assessment; p = .006, t-test, 1 sided; Mean Difference (Final Values) = -0.43, 97.5% CI 1-sided [lower limit -3.26], Standard Error of Mean 1.43; Treatment difference = standard Trauma Focused -CBT - stepped care Trauma Focused-CBT

2. Primary Outcome: Trauma Symptom Checklist for Young Children Posttraumatic Stress Symptoms
Description: as for outcome 1
Time Frame: 6-month Follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 36.84 (11.56) | 36.31 (9.68)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — We planned 0.41 standard deviation (SD) as the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied at 6-month assessment; p = .004, t-test, 1 sided; Mean Difference (Final Values) = -0.53, 97.5% CI 1-sided [lower limit -3.47], Standard Error of Mean 1.49; Treatment difference = standard Trauma Focused -CBT - stepped care Trauma Focused-CBT

3. Primary Outcome: Trauma Symptom Checklist for Young Children Posttraumatic Stress Symptoms
Description: as for outcome 1
Time Frame: 12-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 35.05 (8.26) | 34.92 (9.14)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Based on the actual randomization of 183 participants (SC-TF-CBT=91; standard TF-CBT=92), we had more than 80% power to show that SC-TF-CBT is at least as effective as standard TF-CBT with alpha of .05 and a non-inferior margin of 0.41 standard deviation units; Test type: Non-Inferiority — We planned 0.41standard deviation as the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied 12-month assessment; p = .001, t-test, 1 sided; Mean Difference (Final Values) = -0.13, 97.5% CI 1-sided [lower limit -2.50], Standard Error of Mean 1.20; Treatment difference = standard TF-CBT - stepped care TF-CBT

4. Primary Outcome: Child Sheehan Disability Scale Parent Version
Description: The Child Sheehan Disability Scale is a caregiver report to measure childhood impairment. The change in the impairment scores will be used to measure change in impairment.Scores range from 0 to 50 with higher scores indicating greater impairment.
Time Frame: Post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 12.03 (16.36) | 12.82 (13.28)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — We planned 0.41 standard deviation as the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied at post assessment; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 0.79, 97.5% CI 1-sided [lower limit -2.94], Standard Error of Mean 1.89; Treatment difference = standard TF-CBT - stepped care TF-CBT

5. Primary Outcome: Child Sheehan Disability Scale Parent Version
Description: as for outcome 4
Time Frame: 6-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 13.23 (16.23) | 11.33 (12.93)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — We planned 0.41 standard deviation as the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied at 6-month assessment; p = .044, t-test, 1 sided; Mean Difference (Final Values) = -1.89, 97.5% CI 1-sided [lower limit -6.33], Standard Error of Mean 2.25; Treatment difference = standard TF-CBT - stepped care TF-CBT

6. Primary Outcome: Child Sheehan Disability Scale Parent Version
Description: as for outcome 4
Time Frame: 12-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 7.88 (12.07) | 8.25 (11.38)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — We planned 0.41 standard deviation as the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied at 12-month assessment; p = 0.002, t-test, 1 sided; Mean Difference (Final Values) = 0.38, 97.5% CI 1-sided [lower limit -3.07], Standard Error of Mean 1.75; Treatment difference = standard TF-CBT - stepped care TF-CBT

7. Secondary Outcome: Child Behavior Checklist Internalizing Symptoms
Description: Changes in T scores in internalizing symptoms. T scores may range from 33 to 100 with higher T scores indicating greater internalizing symptoms.
Time Frame: Post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 45.68 (10.42) | 44.62 (10.53)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.016, t-test, 1 sided; Mean Difference (Final Values) = -1.06, 97.5% CI 1-sided [lower limit -4.06], Standard Error of Mean 1.52; Treatment difference = standard TF-CBT - stepped care TF-CBT

8. Secondary Outcome: Child Behavior Checklist Internalizing Symptoms
Description: as for outcome 7
Time Frame: 6-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 47.17 (12.33) | 46.93 (12.52)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.003, t-test, 1 sided; Mean Difference (Final Values) = -0.23, 97.5% CI 1-sided [lower limit -3.72], Standard Error of Mean 1.77; Treatment difference = standard TF-CBT - stepped care TF-CBT

9. Secondary Outcome: Child Behavior Checklist Internalizing Symptoms
Description: as for outcome 7
Time Frame: 12-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 45.71 (12.46) | 45.56 (12.39)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — We planned 0.41 standard deviation the non-inferiority margin (which is less than half of the effect size) for the one-side testing. Non-inferiority analysis with alpha 2.5% was applied at 12-month assessment; p = 0.007, t-test, 1 sided; Mean Difference (Final Values) = -0.16, 97.5% CI 1-sided [lower limit -3.89], Standard Error of Mean 1.89; Treatment difference = standard TF-CBT - stepped care TF-CBT

10. Secondary Outcome: Child Behavior Checklist Externalizing Symptoms
Description: Changes in T scores in externalizing symptoms. T scores range from 33 to 100 with higher T scores indicating greater externalizing problems.
Time Frame: Post treatment
Population: Intent to treat population (ITT: all participants assigned to stepped care TF-CBT and standard TF-CBT). Multiple imputation was applied for ITT analysis, with ten imputations generated at item level and individual level.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 47.41 (12.00) | 46.40 (11.30)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.008, t-test, 1 sided; Mean Difference (Final Values) = -1.01, 97.5% CI 1-sided [lower limit -4.24], Standard Error of Mean 1.64; Treatment difference = standard TF-CBT - stepped care TF-CBT

11. Secondary Outcome: Child Behavior Checklist Externalizing Symptoms
Description: as for outcome 10
Time Frame: 6-month follow up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 49.76 (12.52) | 48.40 (12.47)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.015, t-test, 1 sided; Mean Difference (Final Values) = -1.36, 97.5% CI 1-sided [lower limit -4.88], Standard Error of Mean 1.78; Treatment difference = standard TF-CBT - stepped care TF-CBT

12. Secondary Outcome: Child Behavior Checklist Externalizing Symptoms
Description: as for outcome 10
Time Frame: 12-month follow up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 46.92 (14.82) | 45.17 (12.63)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.024, t-test, 1 sided; Mean Difference (Final Values) = -1.75, 97.5% CI 1-sided [lower limit -5.68], Standard Error of Mean 1.99; Treatment difference = standard TF-CBT - stepped care TF-CBT

13. Secondary Outcome: Clinical Global Impression-Severity (CGI-S)
Description: The CGI-S is a widely used 7-point rating of severity of psychopathology including. impairment (0=no illness, 6=extremely severe). Changes in ratings will be used to measure change in severity.
Time Frame: Post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 1.66 (1.46) | 1.66 (1.52)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.001, t-test, 1 sided; Mean Difference (Final Values) = 0.00, 97.5% CI 1-sided [lower limit -0.39], Standard Error of Mean 0.20; Treatment difference = standard TF-CBT - stepped care TF-CBT

14. Secondary Outcome: Clinical Global Impression-Severity (CGI-S)
Description: as for outcome 13
Time Frame: 6-month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 1.45 (1.47) | 1.41 (1.57)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.003, t-test, 1 sided; Mean Difference (Final Values) = -0.04, 97.5% CI 1-sided [lower limit -0.47], Standard Error of Mean 0.22; Treatment difference = standard TF-CBT - stepped care TF-CBT

15. Secondary Outcome: Clinical Global Impression-Severity (CGI-S)
Description: as for outcome 13
Time Frame: 12-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 1.09 (1.31) | 1.13 (1.25)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 0.03, 97.5% CI 1-sided [lower limit -0.30], Standard Error of Mean 0.17; Treatment difference = standard TF-CBT - stepped care TF-CBT

16. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: The CGI-I modified version, 8-point rating will be used for treatment response. A 1, 2 or 3 will be used to indicate treatment response.
Time Frame: Post treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 2.17 (1.08) | 2.15 (0.98)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.02, 97.5% CI 1-sided [lower limit -0.29], Standard Error of Mean 0.14; Treatment difference = standard TF-CBT - stepped care TF-CBT

17. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: as for outcome 16
Time Frame: 6-month treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 2.16 (1.09) | 2.09 (1.21)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.004, t-test, 1 sided; Mean Difference (Final Values) = -0.07, 97.5% CI 1-sided [lower limit -0.38], Standard Error of Mean 0.16; Treatment difference = standard TF-CBT - stepped care TF-CBT

18. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: as for outcome 16
Time Frame: 12-month follow up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 1.74 (0.83) | 1.78 (0.84)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 0.04, 97.5% CI 1-sided [lower limit -0.19], Standard Error of Mean 0.12; Treatment difference = standard TF-CBT - stepped care TF-CBT

19. Other Pre Specified Outcome: Parenting Stress Scale (PSS)
Description: The PSS scores will be used to measure change in parenting stress. Scores range from 18 to 90 with higher scores indicating higher parenting stress.
Time Frame: Post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 32.46 (10.67) | 32.03 (9.70)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.005, t-test, 1 sided; Mean Difference (Final Values) = -0.43, 97.5% CI 1-sided [lower limit -3.33], Standard Error of Mean 1.47; Treatment difference = standard TF-CBT - stepped care TF-CBT

20. Other Pre Specified Outcome: Parenting Stress Scale (PSS)
Description: as for outcome 19
Time Frame: 6-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 33.77 (13.42) | 32.30 (10.51)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.028, t-test, 1 sided; Mean Difference (Final Values) = -1.47, 97.5% CI 1-sided [lower limit -4.99], Standard Error of Mean 1.78; Treatment difference = standard TF-CBT - stepped care TF-CBT

21. Other Pre Specified Outcome: Parenting Stress Scale (PSS)
Description: as for outcome 19
Time Frame: 12-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 32.26 (11.20) | 31.82 (10.43)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.009, t-test, 1 sided; Mean Difference (Final Values) = -0.44, 97.5% CI 1-sided [lower limit -3.64], Standard Error of Mean 1.62; Treatment difference = standard TF-CBT - stepped care TF-CBT

22. Other Pre Specified Outcome: Depression, Anxiety and Stress Scale (Short Form)- Depression Subscale
Description: The depression subscale self-report will be used to measure change in parent depression, Scores range from 0 to 42 with higher scores indicating higher depressive symptoms.
Time Frame: Post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 5.06 (6.97) | 4.00 (5.40)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.006, t-test, 1 sided; Mean Difference (Final Values) = -1.05, 97.5% CI 1-sided [lower limit -2.82], Standard Error of Mean 0.90; Treatment difference = standard TF-CBT - stepped care TF-CBT

23. Other Pre Specified Outcome: Depression, Anxiety and Stress Scale (Short Form)- Depression Subscale
Description: as for outcome 22
Time Frame: 6-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 4.64 (6.69) | 4.07 (6.00)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.57, 97.5% CI 1-sided [lower limit -2.31], Standard Error of Mean 0.88; Treatment difference = standard TF-CBT - stepped care TF-CBT

24. Other Pre Specified Outcome: Depression, Anxiety and Stress Scale (Short Form)- Depression Subscale
Description: as for outcome 22
Time Frame: 12-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 4.18 (5.66) | 4.39 (5.62)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 1 sided; Median Difference (Final Values) = 0.21, 97.5% CI 1-sided [lower limit -1.43], Standard Error of Mean 0.83; Treatment difference = standard TF-CBT - stepped care TF-CBT

25. Other Pre Specified Outcome: The PTSD Checklist-Civilian (PCL-C)
Description: The PCL-C will be used to measure change in parent self-report of PTSD symptom severity. Scores range from 0 to 80 with higher scores indicating greater posttraumatic stress symptoms.
Time Frame: Post treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 13.40 (15.82) | 12.63 (15.87)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — For the non-inferiority margin for the PCL-5, the clinically significant change threshold is 10 points although adult PTSD trials have used -5 to -10 points. We used -8.8 as the margin which was based on an expert panel and prior studies with adults. Non-inferiority analysis with alpha 2.5% was applied at post assessment; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.77, 97.5% CI 1-sided [lower limit -5.04], Standard Error of Mean 2.16; Treatment difference = standard TF-CBT - stepped care TF-CBT

26. Other Pre Specified Outcome: The PTSD Checklist-Civilian (PCL-C)
Description: as for outcome 25
Time Frame: 6-month follow up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 14.67 (17.78) | 12.27 (14.35)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — For the non-inferiority margin for the PCL-5, the clinically significant change threshold is 10 points although adult PTSD trials have used -5 to -10 points. We used -8.8 as the margin which was based on an expert panel and prior studies with adults. Non-inferiority analysis with alpha 2.5% was applied at 6-month assessment; p = 0.003, t-test, 1 sided; Mean Difference (Final Values) = -2.40, 97.5% CI 1-sided [lower limit -6.87], Standard Error of Mean 2.27; Treatment difference = standard TF-CBT - stepped care TF-CBT

27. Other Pre Specified Outcome: The PTSD Checklist-Civilian (PCL-C)
Description: as for outcome 25
Time Frame: 12-month follow up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
Number analyzed (Participants) | 91 | 92
score on a scale | 13.51 (15.25) | 11.78 (13.77)
Statistical Analysis 1: Comparison: Stepped Care TF-CBT vs Standard TF-CBT; Test type: Non-Inferiority — For the non-inferiority margin for the PCL-5, the clinically significant change threshold is 10 points although adult PTSD trials have used -5 to -10 points. We used -8.8 as the margin which was based on an expert panel and prior studies with adults.Non-inferiority analysis with alpha 2.5% was applied at 12-month assessment; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -1.74, 97.5% CI 1-sided [lower limit -5.80], Standard Error of Mean 2.06; Treatment difference = standard TF-CBT - stepped care TF-CBT

ADVERSE EVENTS:
Time Frame: From enrollment to the end of the the 12 month post treatment follow-up assessment (approximately 1 year, 4 months). Assessed every visit from enrollment to the end of the 12 month post treatment follow up assessment.
Groups:
- Stepped Care TF-CBT: Participants (parents/guardian and children) received Step One which is a parent-led therapist-assisted treatment: 3 therapist-led sessions along with 11 parent-child meetings using a parent-child workbook. Children who do not meet responder status will receive Step Two: 9 therapist-directed sessions of TF-CBT. Two as needed sessions could be provided.
- Standard TF-CBT: Participants (parents/guardians and children) received therapist-led trauma-focused cognitive behavioral therapy (TF-CBT). Two as needed sessions could be provided.
Arm/Group | Stepped Care TF-CBT | Standard TF-CBT
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/184
Serious Adverse Events (participants affected / at risk) | 19/182 | 29/184
Other Adverse Events (participants affected / at risk) | 9/182 | 16/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stepped Care TF-CBT (N=182) | Standard TF-CBT (N=184)
Child abuse report (children) (Social circumstances) | 12 (16) | 15 (19) — A child abuse report was made to authorities if there was reasonable cause to suspect child abuse, and it had not already been reported. Query was made to assess if abuse was reported.
Hospitalized due to psychiatric crisis and for evaluation (children) (Psychiatric disorders) | 2 (2) | 2 (7) — For children: Hospitalized for mental health. All child hospitalizations occured after treatment and before the last 12 month assessment. Interview was used to asses for hospitalizations.
Heart surgery due to chronic condition (children) (Cardiac disorders) | 0 (0) | 1 (1) — For children: Heart surgery. Surgery was planned and child was able to complete study treatment.
Hospitalized due to gastrointestinal issues (children) (Gastrointestinal disorders) | 1 (1) | 0 (0) — For children: Hospitalized due to gastrointestinal issues. Child had pending diagnosis of Crohn's disease. Occured between post-treatment and 12 month follow-up assessment.
Hospitalized due to virus (children) (Infections and infestations) | 1 (1) | 0 (0) — For children: Admitted to the emergency room due to a virus
Suicidal ideation (children) (Psychiatric disorders) | 3 (3) | 6 (7) — For children: Suicidal ideation. A structured assessment was used to assess for suicidal ideation.
Hospitalized due to prior condition (parents/guardians) (General disorders) | 0 (0) | 4 (4) — For parents/guardians: Hospitalized for prior condition.
Hospitalized due to meningitis (parents/guardians) (Infections and infestations) | 0 (0) | 1 (1) — For parents/guardians: Hospitalized due to meningitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stepped Care TF-CBT (N=182) | Standard TF-CBT (N=184)
Worsening of posttraumatic stress symptoms (children) (Psychiatric disorders) | 9 (10) | 16 (26) — For Children: Parents, children ages 7-12, therapists, evaluators rated change in child's posttraumatic stress symptoms since the first assessment. Three minimally worse ratings, or much worse, or very much worse were considered as worsening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT02537678/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form Parent (2019-12-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02537678/ICF_001.pdf
  • Informed Consent Form: Informed Assent Forms for Children (2019-12-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02537678/ICF_002.pdf